CLINICAL TRIAL: NCT00002576
Title: A RANDOMIZED PROSPECTIVE TRIAL OF CHOP VERSUS MCOP IN ELDERLY PATIENTS WITH INTERMEDIATE AND HIGH GRADE NON-HODGKIN'S LYMPHOMA (AGED 65 YEARS AND OVER)
Brief Title: Combination Chemotherapy in Treating Older Patients With Intermediate- or High-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CRC-TU-NH3003; CDR0000063660 (Registry Identifier: PDQ (Physician Data Query)); EU-93028; ISRCTN39268693 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-05

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage II adult lymphoblastic lymphoma; stage II adult Burkitt lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Mitoxantrone; Prednisolone; Vincristine

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: mitoxantrone hydrochloride
Drug: prednisolone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy consisting of cyclophosphamide, vincristine, and prednisolone, with either mitoxantrone or doxorubicin in treating patients with intermediate- or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the treatment-related neurologic and hematologic toxicities of patients aged 65 years and over with intermediate- or high-grade non-Hodgkin's lymphoma randomized to CHOP (cyclophosphamide, doxorubicin, vincristine, prednisolone) vs. MCOP (mitoxantrone, cyclophosphamide, vincristine, prednisolone). II. Compare the survival rate in these patients.

OUTLINE: Randomized study. The following acronyms are used: CHOP CTX/DOX/VCR/PRDL CTX Cyclophosphamide, NSC-26271 DHAD Mitoxantrone, NSC-301739 DOX Doxorubicin, NSC-123127 MCOP DHAD/CTX/VCR/PRDL PRDL Prednisolone, NSC-9900 VCR Vincristine, NSC-67574 Arm I: 4-Drug Combination Chemotherapy. CHOP. Arm II: 4-Drug Combination Chemotherapy. MCOP.

PROJECTED ACCRUAL: A total of 200 patients will be entered over approximately 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed intermediate- or high-grade non- Hodgkin's lymphoma of the following types: Diffuse centroblastic Diffuse immunoblastic B- and T-cell lymphoblastic Peripheral T-cell (mixed or large cell) and Ki-1 No Stage IA (nonbulky) disease suitable for radiotherapy alone

PATIENT CHARACTERISTICS: Age: 65 and over Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No severe ischemic heart disease No cardiomyopathy that would restrict doxorubicin use Other: No other serious medical conditions that would affect treatment outcome No prior malignancy except: Nonmelanomatous skin cancer Adequately treated in situ cervical cancer Sufficiently fit to receive treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1992-11; Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Michael Bessell, MD, PhD, FRCP, FRCR, Study Chair — Nottingham City Hospital
Locations (1):
- Nottingham City Hospital NHS Trust, Nottingham, England, United Kingdom

REFERENCES:
- [Derived] Sattler FR, Mert M, Sankaranarayanan I, Mack WJ, Galle-Treger L, Gonzalez E, Baronikian L, Lee K, Jahani PS, Hodis HN, Dieli-Conwright C, Akbari O. Feasibility of quantifying change in immune white cells in abdominal adipose tissue in response to an immune modulator in clinical obesity. PLoS One. 2020 Sep 3;15(9):e0237496. doi: 10.1371/journal.pone.0237496. eCollection 2020. PMID 32881912